CLINICAL TRIAL: NCT06392503
Title: Establishment of Noninvasive Diagnosis Model for High-risk Varices in Cirrhosis Patients Based on iLivTouch
Brief Title: Noninvasive Diagnosis Model for High-risk Varices in Cirrhosis
Acronym: NID-HRV
Status: Recruiting | Type: Observational
Sponsor: Beijing 302 Hospital (Other)
Collaborators: Qianfoshan Hospital (Other); First Hospital of China Medical University (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Second Hospital of Jilin University (Other); Shengjing Hospital (Other); The Affiliated Hospital Of Guizhou Medical University (Other); The First Hospital of Yulin (Unknown); LanZhou University (Other); Chengdu Third People's Hospital (Unknown); Tianjin Third Central Hospital (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); People's Hospital of Lixin County (Unknown); The Fourth People's Hospital of Qinghai Province (Other); The Fourth People's Hospital of Nanning (Other); The Third People's Hospital of Taiyuan (Other); Central Hospital of Huludao (Unknown); Jixi Infectious Diseases Hospital (Unknown); First Affiliated Hospital of Jiamusi University (Unknown); Benxi Sixth People's Hospital (Unknown); Yuncheng Central Hospital (Other); The First People's Hospital of Zigong City, Sichuan Province (Unknown); Second Affiliated Hospital of Guangzhou Medical University (Other); Ruikang Affiliated Hospital of Guangxi University of Chinese Medicine (Unknown); Guilin People's Hospital (Unknown); Tianjin Binhai New Area Dagang Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: KY-2023-10-59-1
Record Dates: First submitted 2024-04-26; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-03

CONDITIONS: Varices; Liver Cirrhosis
Keywords: diagnostic model; high risk varices; iLivTouch
MeSH Terms: conditions — Varicose Veins; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- retrospective cohort group: patients before the study started
  Interventions: Diagnostic Test: different diagnostic models
- prospective cohort group: spatients after the study started
  Interventions: Diagnostic Test: different diagnostic models

INTERVENTIONS:
Diagnostic Test: different diagnostic models — the patients were screened by different diagnostic models

SUMMARY:
This is an observational ambispective cohort study to validate the Baveno VI guideline and develop a new diagnostic model to screen high-risk varices (HRV) of liver cirrhosis using iLivTouch.

DETAILED DESCRIPTION:
Esophageal variceal bleeding is a common and fatal complication in patients with liver cirrhosis. The diagnosis of high-risk varices (HRV) traditionally depends on gastroscopy, which is expensive and poorly tolerated with patients. Baveno VI guideline has put forward a HRV screening model based on liver stiffness and platelet count. This is an observational ambispective cohort study. The retrospective cohort is derived from the previous records of the hospital information system, and the prospective cohort is enrolled prospectively at the local research center when participants meet the inclusion criteria. The purpose of this study is to establish a diagnostic model of HRV in patients with liver cirrhosis according to the liver stiffness value measured by iLivTouch and other laboratory indexes, so as to verify the applicability of Baveno VI standard under the condition of iLivTouch and establish a cutoff value that is more suitable for iLivTouch. In addition, this study will try to find some new indexes to further improve the diagnostic efficiency of HRV. The minimum enrolment period is anticipated to be 6 months per center and will be extended if necessary to reach the overall study target.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75;
2. Patients with liver cirrhosis diagnosed by clinical or imaging diagnosis;
3. The interval of iLivTouch and esophagogastroduodenoscopy is no more than 3 months;

Exclusion Criteria:

1. the interval between esophagogastroduodenoscopy and iLivTouch is more than 3 months;
2. any decompensation events (ascites, hepatic encephalopathy or gastroesophageal variceal bleeding) during endoscopy or iLivTouch examination, or during the interval between them;
3. currently taking nonselective beta blocker/ antiplatelet / anticoagulant drugs;
4. hepatocellular carcinoma;
5. after transjugular intrahepatic portosystemic shunt surgery;
6. after liver transplantation.
7. portal-spleen-mesenteric venous thrombosis;
8. patients with splenectomy;
9. BMI ≥ 30;
10. patients with acute active hepatitis or patients with cholestatic hepatitis;
11. IQR/median of liver stiffness measurement > 30%.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with liver cirrhosis diagnosed by clinical or imaging diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
diagnostic performance | at end of the patient enrollment
  sensitivity, specificity, positive predictive value, negative predictive value and accuracy of different diagnostic models

OTHER OUTCOMES:
Endoscopy spared ratio | at end of the patient enrollment
  the percentage of patients spared with endoscopy
HRV missing ratio | at end of the patient enrollment
  the percentage of patients missed with high-risk varices

CONTACTS AND LOCATIONS:
Overall Officials: Fu junliang, Principal Investigator — the Fifth Medical Center, Chinese PLA General Hospital
Locations (1):
- the Fifth Medical Center, Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
After enrollment and data analysis, the study results will be submitted to peer-reviewed journals for publication. Personal information about potential and enrolled participants will be strictly confidential to the public before, during, and after the study.

REFERENCES:
- [Background] Yan Y, Xing X, Wang X, Yang L. Liver stiffness by two-dimensional shear wave elastography for screening high-risk varices in patients with compensated advanced chronic liver disease. Eur Radiol. 2022 Mar;32(3):2078-2088. doi: 10.1007/s00330-021-08280-3. Epub 2021 Oct 29. PMID 34713329
- [Background] de Franchis R; Baveno VI Faculty. Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. J Hepatol. 2015 Sep;63(3):743-52. doi: 10.1016/j.jhep.2015.05.022. Epub 2015 Jun 3. No abstract available. PMID 26047908
- [Background] Augustin S, Pons M, Maurice JB, Bureau C, Stefanescu H, Ney M, Blasco H, Procopet B, Tsochatzis E, Westbrook RH, Bosch J, Berzigotti A, Abraldes JG, Genesca J. Expanding the Baveno VI criteria for the screening of varices in patients with compensated advanced chronic liver disease. Hepatology. 2017 Dec;66(6):1980-1988. doi: 10.1002/hep.29363. Epub 2017 Oct 30. PMID 28696510
- [Background] Wang H, Wen B, Chang X, Wu Q, Wen W, Zhou F, Guo Y, Ji Y, Gu Y, Lai Q, He Q, Li J, Chen J, Hou J. Baveno VI criteria and spleen stiffness measurement rule out high-risk varices in virally suppressed HBV-related cirrhosis. J Hepatol. 2021 Mar;74(3):584-592. doi: 10.1016/j.jhep.2020.09.034. Epub 2020 Oct 8. PMID 33039403
- [Background] de Franchis R, Bosch J, Garcia-Tsao G, Reiberger T, Ripoll C; Baveno VII Faculty. Baveno VII - Renewing consensus in portal hypertension. J Hepatol. 2022 Apr;76(4):959-974. doi: 10.1016/j.jhep.2021.12.022. Epub 2021 Dec 30. PMID 35120736
- [Background] Zhang X, Song J, Zhang Y, Wen B, Dai L, Xi R, Wu Q, Li Y, Luo X, Lan X, He Q, Luo W, Lai Q, Ji Y, Zhou L, Qi T, Liu M, Zhou F, Wen W, Li H, Liu Z, Chen Y, Zhu Y, Li J, Huang J, Cheng X, Tu M, Hou J, Wang H, Chen J. Baveno VII algorithm outperformed other models in ruling out high-risk varices in individuals with HBV-related cirrhosis. J Hepatol. 2023 Mar;78(3):574-583. doi: 10.1016/j.jhep.2022.10.030. Epub 2022 Nov 7. PMID 36356684
- [Background] Ng YZ, Lai LL, Wong SW, Mohamad SY, Chuah KH, Chan WK. Attenuation parameter and liver stiffness measurement using FibroTouch vs Fibroscan in patients with chronic liver disease. PLoS One. 2021 May 3;16(5):e0250300. doi: 10.1371/journal.pone.0250300. eCollection 2021. PMID 33939744
- [Background] Ou X, Wang X, Wu X, Kong Y, Duan W, Zhou J, Sun D, Wang Y, You H, Jia J. [Comparison of FibroTouch and FibroScan for the assessment of fibrosis in chronic hepatitis B patients]. Zhonghua Gan Zang Bing Za Zhi. 2015 Feb;23(2):103-6. doi: 10.3760/cma.j.issn.1007-3418.2015.02.006. Chinese. PMID 25880975
- [Background] Zeng J, Sun WL, Chen GY, Pan Q, Yan SY, Sun C, Xu ZJ, Fan JG. [Efficiency of FibroScan and FibroTouch in liver stiffness measurement and fat quantification: a comparative analysis]. Zhonghua Gan Zang Bing Za Zhi. 2016 Sep 20;24(9):652-658. doi: 10.3760/cma.j.issn.1007-3418.2016.09.004. Chinese. PMID 27788720
- [Background] Colecchia A, Ravaioli F, Marasco G, Colli A, Dajti E, Di Biase AR, Bacchi Reggiani ML, Berzigotti A, Pinzani M, Festi D. A combined model based on spleen stiffness measurement and Baveno VI criteria to rule out high-risk varices in advanced chronic liver disease. J Hepatol. 2018 Aug;69(2):308-317. doi: 10.1016/j.jhep.2018.04.023. Epub 2018 May 3. PMID 29729368